CLINICAL TRIAL: NCT01061320
Title: Efficacy of Alpha Tocopherol and New Biomarker (Urine NGAL) for Prevention and Early Diagnosis of Contrast-induced Nephropathy in CKD Patients Undergoing Elective Coronary Procedures
Brief Title: Efficacy of Alpha Tocopherol for Prevention of Contrast-induced Nephropathy in Chronic Kidney Disease (CKD) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Thammasat University (Other)
Responsible Party: Adis Tasanarong, Faculty of Medicine, Thammasat University (Rangsit Campus)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTU-I-1-53/52
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-01

CONDITIONS: Contrast Induced Nephropathy
Keywords: Alpha-Tocopherol (Vitamin E); Contrast induced nephropathy; Chronic kidney disease; Coronary procedures
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — alpha-Tocopherol; Tocopherols; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alpha tocopherol (Active Comparator)
  Interventions: Drug: alpha tocopherol
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alpha tocopherol — The patients were assigned to receive oral alpha tocopherol (525 IU) every day start at five day before procedure, in the morning before procedure and 24 hr post-coronary procedure.
  Other Names: Bio-E-vitamin
  Arms: alpha tocopherol
Drug: placebo — The patients were assigned to receive oral placebo every day start at five day before procedure, in the morning before procedure and 24 hr post-coronary procedure.
  Other Names: jelly
  Arms: placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of alpha tocopherol for prevention contrast-induced nephropathy in CKD patients undergoing elective coronary procedures.

DETAILED DESCRIPTION:
Contrast-induced nephropathy (CIN) increases the likelihood of patient morbidity and mortality following coronary procedures. Contrast agents cause an acute deterioration in renal function via the generation of reactive oxygen species. Vitamin E (alpha tocopherol)was demonstrated to be anti-oxidant and anti-inflammation. The present study was designed to evaluate the administration of antioxidant vitamin E (alpha tocopherol) as a means of preventing CIN in these patients.

ELIGIBILITY:
Inclusion Criteria:

* serum creatinine levels > 1.2 mg/dL and baseline creatinine clearance levels < 60 mL/min (as measured in their most recent sample,drawn within 2 months prior to the beginning of the study)

Exclusion Criteria:

* patients with acute kidney injury
* end stage renal disease (requiring dialysis)
* unstable renal function (as evidenced by a change in serum creatinine of > 0.5 mg/dL, or > 25%, within 14 days prior to the study)
* allergy to any of the contrast agents
* mechanical ventilation
* suffered from congestive heart failure, cardiogenic shock or emergent angiography.
* receiving NAC, mannitol, diuretics, theophylline, dopamine, vitamin E or contrast agents within 14 days before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary end-point of this study is the development of CIN in placebo group compared with alpha tocopherol group. | 1 year

SECONDARY OUTCOMES:
The secondary end-point of this study is compare urine NGAL level in CIN patients between both groups. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adis Tasanarong, MD, Principal Investigator — Faculty of Medicine, Thammasat University (Rangsit Campus)
Locations (1):
- Adis Tasanarong, Khlong Luang, Pathumtani, Thailand

REFERENCES:
- [Result] Tasanarong A, Piyayotai D, Thitiarchakul S. Protection of radiocontrast induced nephropathy by vitamin E (alpha tocopherol): a randomized controlled pilot study. J Med Assoc Thai. 2009 Oct;92(10):1273-81. PMID 19845233
- See also: The Nephrology Society of Thailand — http://www.nephrothai.org/